CLINICAL TRIAL: NCT06108258
Title: Newborn Phosphocalcic Metabolism After Intravenous Iron Administration During Pregnancy
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Fanny Schumacher, resident doctor, University Hospital, Geneva
Other Study IDs: 2022-00197
Record Dates: First submitted 2023-10-19; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Iron Induced Hypophosphatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral iron
- IV iron
  Interventions: Drug: IV iron administration

INTERVENTIONS:
Drug: IV iron administration — IV iron administration during pregnancy
  Groups: IV iron

SUMMARY:
Iron deficiency anemia (IDA) is a very common health problem during pregnancy and intravenous (IV) iron substitution has become part of routine management. Recent studies have raised concerns about association of IV iron infusion and development of secondary transitory hypophosphatemia (HP) in adults including pregnant women. The study aimed to evaluate the impact of IV iron administration during pregnancy on newborn's phosphatemia.

The investigators conducted a prospective, single-center, observational study in the Geneva University Hospitals (HUG), from September 2022 to March 2023. Pregnant women treated either with IV iron or with oral iron during pregnancy were included. At delivery, a maternal blood sample to assess hemoglobin, hematocrit, ferritin, phosphate and calcium and an umbilical cord blood sample to assess levels of phosphate and calcium were collected. Difference in demographics and clinical characteristics between the two groups were explored using univariate analyses. Multivariate analyses were performed to test the contribution of IV iron substitution on cord blood phosphatemia and calcemia, considering potential confounding factors. Neonatal HP was defined as a phosphate level lower than 1.3 mmol/L.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy
* Term (>37SA) pregnancy
* Oral or IV iron substitution from second trimester

Exclusion Criteria:

* Multiple pregnancy
* Fetal anomalies
* Preterm birth

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with an uncomplicated term (≥ 37 weeks) single pregnancy who received IV iron or oral iron substitution from the 2nd trimester of pregnancy (>12 weeks of pregnancy) to the day of delivery
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Concentration of cord blood phosphate in neonates | Single timepoint at delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No